CLINICAL TRIAL: NCT01936038
Title: Effectiveness of Upper Airway Toning as Adjuvant Treatment in the Former Period of Adaptation of the Continuous Positive Airway Pressure
Brief Title: Upper Airway Toning for Improve the Compliance of CPAP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fisiolistic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Upper Airway Toning - 001
Record Dates: First submitted 2013-08-24; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: CPAP; Upper Airway Toning; Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): CPAP
  Interventions: Other: CPAP
- EXPERIMENTAL GROUP (Experimental): Upper Airway Toning for Improve the Compliance of CPAP
  Interventions: Other: CPAP; Procedure: Upper Airway Toning for Improve the Compliance of CPAP

INTERVENTIONS:
Other: CPAP — CPAP
Procedure: Upper Airway Toning for Improve the Compliance of CPAP — Upper Airway Toning for Improve the Compliance of CPAP
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The obstructive sleep apnoea/hypopnoea syndrome (OSAHS) is a breathing disorder which happens at night and consists of the interruption of airflow for more than five seconds. His current treatment by continuous positive pressure nocturnal machine (CPAP) is not curative and therefore the level of compliance is key to patient improvement. Many patients don´t tolerate CPAP by the numerous side effects involved. The Upper Airway Toning is a compendium of non-invasive techniques that aim to assist tolerance and compliance with the CPAP. These techniques are: oropharyngeal exercises executed actively by the patient for the muscle toning of the upper airways, electrostimulation of the muscles in the floor of the mouth, correction of the tongue position, nasal and bronchial fogging, execution of respiratory gymnastics, therapy myofascial in the oropharyngeal muscles, manual therapy in the cervical column,and massage in the diaphragm. All the techniques together seek for a greater or lesser impact on the upper airways hypotony, the hypotony of the tongue and the soft palate, the jaw retrognathism, the mouth breathing, the vertebrobasilar syndrome, the gastroesophageal reflux, the excessive accumulation of secretions in the upper and lower airways, the obstructive and restrictive respiratory problems, the sleeping posture, the hypertonia of the diaphragm due to the excess effort in trying to overcome the respiratory obstruction. All these disfunctions will make easier for the patient to show side effects in the use of CPAP. There will be a double-blind randomized controlled study with 110 individuals. One group will follow the conventional medical treatment with CPAP and the other group medical treatment plus Upper Airway Toning. After six months, the mean improvement between the two groups will be compared.

DETAILED DESCRIPTION:
OBJECTIVES

Main objective: To increase the percentage of Nasal Continuous Positive Airway Pressure (nCPAP) compliance.

Secondary objectives:

* To increase the CPAP's tolerance.
* To decrease the CPAP's pressure.
* To decrease the daytime sleepiness.
* To increase the quality of life related to sleep.
* To assess the level of subjective utility of CPAP by the patient.

METHODOLOGY

Type of study: Controlled randomized simple blind study

Randomization of groups

Once the patient is into the study (because s/he has the inclusion criteria and has signed up the informed consent), an opaque envelope is opened in order to know the assigned group.The envelopes are consecutively numbered and the assigned group is randomized through the software.

* Group 1 or control group: 55 subjects undergo the CPAP treatment.
* Group 2 or study group: 55 subjects undergo the CPAP treatment and Upper Airway Toning.

Homogeneity of groups:

Investigators check out the homogeneity of groups in baseline:

Specific features: Neck circumference, presence or lack of nasal clinic, presence or lack of nasal structural alteration, age, gender, weight, height, BMI, smoking habits.

Polysomnographic parameters: Number of apnea, number of hypo-apneas and Apnea Hypopnea Index (AHI).

Symptoms: Presence or lack of severe comorbidities, level of daily hyper-somnolence, presence of insomnia

ELIGIBILITY:
Inclusion Criteria:

* Patients with OSA using CPAP

Exclusion Criteria:

* Neurological Patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
CPAP compliance | 3 months
  nominal variable

SECONDARY OUTCOMES:
Sleep Apnea Quality of Life Index (SAQLI) Test | 3 months
  Test of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Estelle, Principal Investigator — Hospital Universitari General de Catalunya; Anna Bagué, Study Chair — Fisiolístic; Xavier Gironés, Study Chair — Universitat Internacional de Catalunya; Montserrat Girabent, Study Chair — Universitat General de Catalunya; Eduard Estivill, Study Chair — Clínica Dexeus; Francesc Segarra, Study Chair — Hospital Universitari General de Catalunya
Locations (1):
- Fisiolistic, L'Hospitalet de Llobregat, Barcelona, Spain